CLINICAL TRIAL: NCT02647554
Title: A Prospective, Multi-Centre, Double-Blind, Randomized, Placebo-Controlled, Trial of Ulinastatin Treatment in Adult Patients With Sepsis and Septic Shock in China
Brief Title: Ulinastatin Treatment in Adult Patients With Sepsis and Septic Shock in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Techpool Bio-Pharma Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Bin Du, Director of Medical ICU, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UTI-S001
Record Dates: First submitted 2015-12-27; First posted 2016-01-06 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Sepsis; Septic Shock
Keywords: sepsis; septic shock; Ulinastatin; adult; China
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — urinastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ulinastatin group (Experimental): Ulinastain treatment group：400,000 IU ulinastatin will be reconstituted in 10 mL of 0.9% normal saline, and then dissolved in 100 mL of 0.9% normal saline every 8 hours for 10 days in a double-blind fashion.
  Interventions: Drug: ulinastatin
- Placebo group (Placebo Comparator): Placebo control group：Matching with medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ulinastatin — ulinastatin 400,000 IU every 8 hours for 10 days
  Other Names: urinary trypsin inhibitor
  Arms: Ulinastatin group
Drug: Placebo — matching placebo every 8 hours for 10 days
  Arms: Placebo group

SUMMARY:
A Prospective, Multi-Centre, Double-Blind, Randomized, Placebo-Controlled, Trial of Ulinastatin Treatment in Adult Patients with Sepsis and Septic Shock in China

DETAILED DESCRIPTION:
Investigational drug：Ulinastain for Injection

Study title： A Prospective, Multi-Centre, Double-Blind, Randomized, Placebo-Controlled, Trial of Ulinastatin Treatment in Adult Patients with Sepsis and Septic Shock in China

Principal Investigator：Professor Bin Du, Medical Intensive Care Unit, Peking Union Medical College Hospital; Professor Xiangyou Yu, Critical Care Medicine, First Affiliated Hospital, Xinjiang Medical University

Study subjects： Adult patients with sepsis and septic shock will be eligible for inclusion if all of the inclusion criteria are met within 48 hours of meeting criteria of sepsis-3 definition

Study phase： Investigator Initiated Trial(IIT)

Study objectives： The primary objective of the study is to determine whether ulinastatin, compared to placebo, reduces 28-day all-cause mortality in patients with sepsis and septic shock

Study design： Prospective, Multi-Centre, Double-Blind, Randomized, Placebo-Controlled, Clinical Trial

Medication method：

* Ulinastain treatment group： 400,000 IU ulinastatin or matching placebo will be reconstituted in 10 mL of 0.9% normal saline, and then dissolved in 100 mL of 0.9% normal saline every 8 hours for 10 days in a double-blind fashion. Intravenous infusion, The study drug will be infused intravenously over 1 hour.
* Placebo control group：Matching with medication

Course：10 days

Sample size： 348(174 patients of treatment group, 174 patients of control group)

Sites： 15

Primary endpoint：The primary outcome measure for the study is death from all causes at 28-days.

Secondary endpoints:

* Mortality rate at 90-days
* Mortality rate in ICU
* Mortality rate at hospital discharge
* ICU-free days in 28 days
* Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score at 1, 3, 6, 10,14, and 28 days after randomization
* Incidence and duration of supportive care for organ dysfunction including vasoactive agents, invasive or noninvasive mechanical ventilation, continuous renal replacement therapy(CRRT)
* Blood lactate concentration at 1, 3, 6 and 10 days after randomization
* Condition of fluid balance within 10 days after randomization
* High-sensitivity C-reactive protein (hs-CRP), IL-6, IL-10, TNF-α at 1, 3,6 and 10 days after randomization
* ADL level at hospital discharge

Safety endpoints

* adverse events
* serious adverse events
* vital signs, complete blood counts, chemistry, electrocardiograms

ELIGIBILITY:
Inclusion Criteria:Patients will be eligible for inclusion if all of the inclusion criteria are met

1) Sepsis-3 criteria from Society of Critical Care Medicine (SCCM) /European Society of Intensive Care Medicine(ESICM)

1. Suspected or confirmed infection AND
2. Evidence of acute organ dysfunction • in patients not known to have preexisting organ dysfunction (The baseline SOFA score can be assumed to be zero): total SOFA score ≥2 points from 48 hours before infection to 24 hours after infection.

   • in patients known to have preexisting organ dysfunction (The baseline SOFA score can be assumed according to baseline conditions): changes of total SOFA score ≥2 points from 48 hours before infection to 24 hours after infection.

   2）48 hours within diagnosis of sepsis 3）Signed and dated informed consent should be obtained prior to any screening procedures from subjects (or legal representatives). If the subject is unable to provide consent, it could be obtained from legal representatives according to local regulation. Consent from subject should be obtained afterwards when available.

   4） Fertile men or women should agree to use efficient birth control methods during the treatment period and at least 28 days after last dose. Fertile is defined as biologically fertile and sexually active from investigator's view.

   5） Non-childbearing women (meet at least one of following criteria):

   • Past hysterectomy or bilateral oothectomy；

   • Medically confirmed ovarian failure, or menopause (amenorrhea for 12 month or more and with no other pathological or physiological reason)

   Exclusion Criteria:

   1) Age < 18 years, or age>80 years 2) Pregnancy or lactating 3) New York Heart Association Class IV congestive heart failure, nonseptic cardiogenic shock, or uncontrolled acute blood loss 4) Severe, preexisting, parenchymal liver disease with clinically significant portal hypertension, Child-Pugh C stage cirrhosis or acute liver failure 5) Receipt of a solid-organ or bone marrow transplant 6) Advanced pulmonary fibrosis or non invasive ventilation before study entry 7) Myocardial infarction within the previous 3 months 8) Cardiopulmonary resuscitation within 72 hours before study entry 9） Invasive fungal infection or active pulmonary tuberculosis 10) Full-thickness thermal or chemical burn involving 30% or more of body surface area 11) Evidence of significant drug- or disease-induced immunosuppression

   · Evidence of moderate or severe neutropenia, i.e. absolute neutrophil count (ANC) < 1.0 x 10^9/L
   * Administration of high doses of corticosteroids, i.e. doses of > 20 mg/day of prednisone or equivalent, for ≥ 2 weeks immediately prior to evaluation for enrollment. Hydrocortisone at dose ≤ 300 mg/d for treatment of septic shock is acceptable.
   * Immunomodulatory medication (e.g. cyclosporine, azathioprine, OKT3), chemotherapy, or radiation therapy within 2 months before study entry
   * Known HIV seropositivity
   * Any disease sufficiently advanced to suppress resistance to infection
   * Non-remission stage of hematological/lymphoid tumor 12) Previous Xuebijing, thymosin or IVIG Within 2 months before study entry 12) Inability to obtain informed consent or assent 13) Participation in an investigational clinical trial within 6 months of screening 14) Expected survival < 2 months or chronic vegetative state 15) Lack of commitment to full, aggressive, life support 16) History of hypersensitivity to ulinastatin or any excipients or preservatives

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2016-12; Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 28 days
  death from all causes at 28-days

SECONDARY OUTCOMES:
mortality | 90 days
  mortality rate at 90 days
mortality in ICU | through ICU discharge, an average of 14 days
  mortality rate at ICU discharge
mortality rate at hospital discharge | through hospital discharge, an average of 21 days
  mortality rate at hospital discharge
ICU-free days | 28 days
  The time not indwelling in ICU in 28 days
SOFA score | Day 1,3,6,10,14,28 after randomization
  Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score at 1, 3, 6, 10,14, and 28 days after randomization
incidence of supportive care | through ICU discharge, an average of 14 days
  Incidence of supportive care for organ dysfunction including vasoactive agents, invasive or noninvasive mechanical ventilation, continuous renal replacement therapy(CRRT)
duration of supportive care | through ICU discharge, an average of 14 days
  Duration of supportive care for organ dysfunction including vasoactive agents, invasive or noninvasive mechanical ventilation, continuous renal replacement therapy(CRRT)
blood lactate concentration | Day 1,3,6,10 after randomization
  Blood lactate concentration at 1, 3, 6 and 10 days after randomization
fluid balance | through ICU discharge, an average of 10 days
  Condition of fluid balance in ICU after randomization
serum hsCRP | Day 1,3,6,10 after randomization
  High-sensitivity C-reactive protein (hs-CRP) at 1, 3,6 and 10 days after randomization
serum IL-6 | Day 1,3,6,10 after randomization
  IL-6 at 1, 3,6 and 10 days after randomization
serum IL-10 | Day 1,3,6,10 after randomization
  IL-10 at 1, 3,6 and 10 days after randomization
serum TNF-α | Day 1,3,6,10 after randomization
  TNF-α at 1, 3,6 and 10 days after randomization
complete blood counts | Day 1-10, 14, 28 after randomization
  Complete blood counts at 1-10, 14, 28 days after randomization
liver function (alanine aminotransferase, ALT) | Day 1-10, 14, 28 after randomization
  Hepatic (ALT) function tests at 1-10,14 and 28 days after randomization
liver function (Aspartate transaminase, AST) | Day 1-10, 14, 28 after randomization
  Hepatic (AST) function tests at 1-10,14 and 28 days after randomization
liver function (bilirubin) | Day 1-10, 14, 28 after randomization
  Hepatic (bilirubin) function tests at 1-10,14 and 28 days after randomization
respiratory function | Day 1-10, 14, 28 after randomization
  respiratory(PaO2/FiO2) function tests at 1-10,14 and 28 days after randomization
renal function | Day 1-10, 14, 28 after randomization
  renal (creatinine) function tests at 1-10,14 and 28 days after randomization
Activities of daily living (ADL) at hospital discharge | through hospital discharge, an average of 21 days
  Activities of daily living (ADL) level at hospital discharge. This scale is used to assess the patient's ability to run a daily living
adverse events | till 28 days after randomization
  incidence, duration and severity of adverse events
serious adverse events | till 28 days after randomization
  incidence, duration and severity of serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bin Du, MD, Principal Investigator — Peking Union Medical College Hospital, Beijing, China
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chalfin DB, Holbein ME, Fein AM, Carlon GC. Cost-effectiveness of monoclonal antibodies to gram-negative endotoxin in the treatment of gram-negative sepsis in ICU patients. JAMA. 1993 Jan 13;269(2):249-54. PMID 8417245
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Finfer S, Bellomo R, Lipman J, French C, Dobb G, Myburgh J. Adult-population incidence of severe sepsis in Australian and New Zealand intensive care units. Intensive Care Med. 2004 Apr;30(4):589-96. doi: 10.1007/s00134-004-2157-0. Epub 2004 Feb 12. PMID 14963646
- [Background] Padkin A, Goldfrad C, Brady AR, Young D, Black N, Rowan K. Epidemiology of severe sepsis occurring in the first 24 hrs in intensive care units in England, Wales, and Northern Ireland. Crit Care Med. 2003 Sep;31(9):2332-8. doi: 10.1097/01.CCM.0000085141.75513.2B. PMID 14501964
- [Background] Brun-Buisson C, Meshaka P, Pinton P, Vallet B; EPISEPSIS Study Group. EPISEPSIS: a reappraisal of the epidemiology and outcome of severe sepsis in French intensive care units. Intensive Care Med. 2004 Apr;30(4):580-8. doi: 10.1007/s00134-003-2121-4. Epub 2004 Mar 2. PMID 14997295
- [Background] Cheng B, Xie G, Yao S, Wu X, Guo Q, Gu M, Fang Q, Xu Q, Wang D, Jin Y, Yuan S, Wang J, Du Z, Sun Y, Fang X. Epidemiology of severe sepsis in critically ill surgical patients in ten university hospitals in China. Crit Care Med. 2007 Nov;35(11):2538-46. doi: 10.1097/01.CCM.0000284492.30800.00. PMID 17828034
- [Background] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Nov 21;369(21):2063. doi: 10.1056/NEJMc1312359. No abstract available. PMID 24256390
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] Christaki E, Anyfanti P, Opal SM. Immunomodulatory therapy for sepsis: an update. Expert Rev Anti Infect Ther. 2011 Nov;9(11):1013-33. doi: 10.1586/eri.11.122. PMID 22029521
- [Background] Sharony R, Yu PJ, Park J, Galloway AC, Mignatti P, Pintucci G. Protein targets of inflammatory serine proteases and cardiovascular disease. J Inflamm (Lond). 2010 Aug 30;7:45. doi: 10.1186/1476-9255-7-45. PMID 20804552
- [Background] Inoue K, Takano H, Yanagisawa R, Yoshikawa T. Protective effects of urinary trypsin inhibitor on systemic inflammatory response induced by lipopolysaccharide. J Clin Biochem Nutr. 2008 Nov;43(3):139-42. doi: 10.3164/jcbn.2008059. Epub 2008 Oct 31. PMID 19015747
- [Background] Huang N, Wang F, Wang Y, Hou J, Li J, Deng X. Ulinastatin improves survival of septic mice by suppressing inflammatory response and lymphocyte apoptosis. J Surg Res. 2013 Jun 15;182(2):296-302. doi: 10.1016/j.jss.2012.10.043. Epub 2012 Nov 9. PMID 23158408
- [Background] Shao YM, Zhang LQ, Deng LH, Yao HG. [Clinical study on effects of ulinastatin on patients with systemic inflammatory response syndrome]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2005 Apr;17(4):228-30. Chinese. PMID 15836828
- [Background] Karnad DR, Bhadade R, Verma PK, Moulick ND, Daga MK, Chafekar ND, Iyer S. Intravenous administration of ulinastatin (human urinary trypsin inhibitor) in severe sepsis: a multicenter randomized controlled study. Intensive Care Med. 2014 Jun;40(6):830-8. doi: 10.1007/s00134-014-3278-8. Epub 2014 Apr 16. PMID 24737258
- [Background] Yuhara H, Ogawa M, Kawaguchi Y, Igarashi M, Shimosegawa T, Mine T. Pharmacologic prophylaxis of post-endoscopic retrograde cholangiopancreatography pancreatitis: protease inhibitors and NSAIDs in a meta-analysis. J Gastroenterol. 2014 Mar;49(3):388-99. doi: 10.1007/s00535-013-0834-x. Epub 2013 May 30. PMID 23720090
- [Derived] Jiang W, Yu X, Sun T, Chai Y, Chang P, Chen Z, Pan J, Peng Z, Wang R, Wang X, Xu Y, Yu L, Zheng Q, Du B; China Critical Care Clinical Trials Group (CCCCTG). ADJunctive Ulinastatin in Sepsis Treatment in China (ADJUST study): study protocol for a randomized controlled trial. Trials. 2018 Feb 21;19(1):133. doi: 10.1186/s13063-018-2513-y. PMID 29467017
- Available data/document: Study Protocol — http://pan.baidu.com/s/1eQJUJDK